CLINICAL TRIAL: NCT02234544
Title: Estudo clínico Randomizado, Controlado e Duplo-cego do Impacto da inibição de um Transportador de Membrana do Colesterol na absorção da Vitamina D
Brief Title: Effect of an Inhibitor of Cholesterol Absorption on Vitamin D Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Mariana Costa Silva, MD, MSc, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 14-0378
Record Dates: First submitted 2014-08-31; First posted 2014-09-09 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; absorption; ezetimibe
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ezetimibe; Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + Cholecalciferol (Placebo Comparator): The groups will be randomized to ezetimibe or placebo. All participants will receive orally a cholecalciferol capsule.
  Interventions: Drug: Cholecalciferol; Other: Placebo
- Ezetimibe + Cholecalciferol (Active Comparator): The groups will be randomized to ezetimibe or placebo. All participants will receive orally a cholecalciferol capsule.
  Interventions: Drug: Ezetimibe; Drug: Cholecalciferol

INTERVENTIONS:
Drug: Ezetimibe — The groups will be randomized to ezetimibe 10 mg for 5 days or placebo. On the fifth day, they should came after an overnight fast for blood tests collection [25(OH)D, PTH, calcium, albumin]. Next, all participants will receive orally a cholecalciferol 50,000 IU capsule and a snack containing 15g of fat. Participants will return 14 days after that for a second blood test.
  Arms: Ezetimibe + Cholecalciferol
Drug: Cholecalciferol — All participants will receive orally a cholecalciferol 50,000 IU capsule and a snack containing 15g of fat. Participants will return 14 days after that for a second blood test.
  Other Names: Vitamin D
Other: Placebo — The groups will be randomized to ezetimibe 10 mg for 5 days or placebo. On the fifth day, they should came after an overnight fast for blood tests collection [25(OH)D, PTH, calcium, albumin]. Next, all participants will receive orally a cholecalciferol 50,000 IU capsule and a snack containing 15g of fat. Participants will return 14 days after that for a second blood test.
  Arms: Placebo + Cholecalciferol

SUMMARY:
Double-blind randomized controlled trial to evaluate the serum levels of 25(OH)D after a single oral dose of cholecalciferol 50,000 IU plus ezetimibe or placebo.

Differences between the serum levels of 25(OH)D in response to cholecalciferol plus ezetimibe compared to cholecalciferol plus placebo.

DETAILED DESCRIPTION:
Objectives: To evaluate the serum levels of 25(OH)D after a single oral dose of cholecalciferol 50,000 IU plus ezetimibe or placebo.

Experimental design: Double-blind randomized controlled trial. Research location: Porto Alegre Clinical Hospital (HCPA), RS, Brazil. Participants: Medical residents of the HCPA. Intervention: The groups will be randomized to ezetimibe 10 mg for 5 days or placebo. On the fifth day, they should came after an overnight fast for blood tests collection [25(OH)D, PTH, calcium, albumin]. Next, all participants will receive orally a cholecalciferol 50,000 IU capsule and a snack containing 15g of fat. Participants will return 14 days after that for a second blood test.

Statistical Analysis: Paired samples t-test or Wilcoxon signed rank-test will be used for comparing variables in two distinct moments (before cholecalciferol and 14 days after). The correlation between the numerical variables will be evaluated by the Spearman's correlation coefficient. A p value of less than 0.05 was considered statistically significant.

Expected results: Differences between the serum levels of 25(OH)D in response to cholecalciferol plus ezetimibe compared to cholecalciferol plus placebo.

Cost/benefit of the project: This is a low budget and minimal risks study that will contribute to a better understanding of the absorptive process of vitamin D and the effect of ezetimibe on its absorption.

ELIGIBILITY:
Inclusion Criteria:

* Medical students of the HCPA

Exclusion Criteria:

* Body mass index >+ 25 or < 18.5 kg/m2
* Known liver, kidney or endocrine disease
* Known malabsorption
* Use of supplements of calcium and/or vitamin Danticonvulsants, barbiturates, or glucocorticoids
* Travel outside the Brazilian south region during the previous 120 days

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D | up to 24 months
  The groups will be randomized to ezetimibe 10 mg for 5 days or placebo. On the fifth day, they should came after an overnight fast for blood tests collection [25(OH)D, PTH, calcium, albumin]. Next, all participants will receive orally a cholecalciferol 50,000 IU capsule and a snack containing 15g of fat. Participants will return 14 days after that for a second blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Silva MC, Faulhauber GAM, Leite EN, Goulart KR, Ramirez JMA, Cocolichio FM, Furlanetto TW. Impact of a cholesterol membrane transporter's inhibition on vitamin D absorption: A double-blind randomized placebo-controlled study. Bone. 2015 Dec;81:338-342. doi: 10.1016/j.bone.2015.07.022. Epub 2015 Jul 21. PMID 26208795